CLINICAL TRIAL: NCT06288880
Title: The Impact of Earthquake Trauma on Compassion Fatigue Among Nurses Working in Emergency Services After the February 6th Kahramanmaraş (Turkey) Earthquakes: A Multicenter Cross-Sectional Study
Brief Title: Impact of Earthquake Trauma on Nurses' Compassion Fatigue: A Study From Kahramanmaraş, Turkey
Status: Not yet recruiting | Type: Observational
Sponsor: Kilis 7 Aralik University (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, İslam Elagöz, Researcher Asisstan, Kilis 7 Aralik University
Other Study IDs: kilis_4
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Earthquake; Compassion Fatigue
Keywords: Earthquake Trauma; Compassion Fatigue; Emergency Service Nurses; Post-Traumatic Stress Disorder (PTSD); Secondary Traumatic Stress Disorder; Kahramanmaraş Earthquakes; Psychological Impact; Healthcare Professionals; Disaster Response; Trauma Care
MeSH Terms: conditions — Compassion Fatigue; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the impact of earthquake trauma on compassion fatigue among nurses working in emergency services following the devastating earthquakes on 6 February 2023, in Kahramanmaraş, Turkey. These earthquakes, with magnitudes of approximately 7.7 and 7.6, affected 11 provinces and resulted in over 50,000 deaths and 100,000 injuries, placing emergency service nurses at the forefront of dealing with the aftermath and trauma. The concept of compassion fatigue, characterised by a reduced capacity for empathy after repeated exposure to traumatic events, is a significant concern for nurses who have been directly involved in the care of earthquake victims. This study aims to explore the extent of earthquake trauma and compassion fatigue among these nurses, examining the relationship between these two conditions and their long-term effects. Given the limited research on post-traumatic stress disorder and compassion fatigue among emergency service nurses, this study seeks to contribute valuable insights into the psychological impacts of disaster response on healthcare professionals. The hypotheses tested aim to better understand the risks and psychological burdens faced by nurses in the wake of such natural disasters.

DETAILED DESCRIPTION:
On 6 February 2023, two earthquakes with magnitudes of approximately 7.7 Mw and 7.6 Mw occurred at 04:17 and 13:24 local time, centred in Kahramanmaraş, Turkey. These earthquakes affected a wide geographical area encompassing 11 provinces of Turkey (Kahramanmaraş, Hatay, Adıyaman, Gaziantep, Malatya, Kilis, Diyarbakır, Adana, Osmaniye, Şanlıurfa, and Elâzığ), leading to significant destruction. As a result of this disaster, more than 50,000 people lost their lives, and over 100,000 were injured. Emergency service nurses, in particular, were at the forefront of this catastrophe, witnessing moments of intense trauma. Nurses working in emergency services had to care for patients with open wounds, closed and open fractures, vascular injuries, compartment syndrome, crush syndrome, amputations, and more. Such traumatic experiences have caused emergency service nurses to suffer from earthquake trauma to a greater extent. Consequently, stress disorders following trauma caused by the earthquake are a serious and common condition among emergency service nurses working in the earthquake zone.

Another issue encountered by emergency service nurses serving people exposed to trauma during the earthquake is compassion fatigue. Compassion fatigue, a term coined by Joinson (1992) to describe the state of burnout experienced by nurses working in emergency services, is known in the international literature as "compassion fatigue" and is referred to as "şefkat yorgunluğu," "merhamet yorgunluğu," and "eş duyum yorgunluğu" in Turkey. Compassion fatigue is also known as secondary traumatic stress disorder, secondary victimisation, and indirect trauma. It is characterised by a reduced capacity for empathy following repeated exposure to traumatic situations experienced by others.

Exposure to such stressful and traumatic workplace events can lead to burnout, post-traumatic stress disorders, depression, anxiety, and other mental health issues related to trau. A systematic review reported significant symptoms of post-traumatic stress disorder and psychological distress among nurses working in the earthquake zone. Another study showed that 25% of emergency service nurses experienced severe depression and sleep disorders, with their anxiety levels being higher than those of nurses working in other unit. A systematic review covering the years 1989-2019 reported that 25.8% of emergency service nurses showed symptoms of post-traumatic stress disorder following experienced traumas. Looking at related studies on compassion fatigue, it is indicated that professionals exposed to trauma victims, such as emergency service workers, disaster workers, emergency service nurses, doctors, and social workers, are at a high risk of compassion fatigue.

In light of the current information, it is clearer that nurses serving in emergency services are at high risk for earthquake trauma and compassion fatigue. Especially in disaster situations like earthquakes, exposure to such conditions reaches its peak, significantly increasing this risk. It has been shown that nurses experiencing psychological health problems may have a decrease in care quality and an increased likelihood of making medical errors. Therefore, determining the level of earthquake trauma and compassion fatigue symptoms among nurses exposed to the 6 February Kahramanmaraş earthquakes, identifying the relationship between these two conditions, and determining their long-term effects will make significant contributions to the effective and efficient implementation of rehabilitation efforts. Given the limited number of studies examining post-traumatic stress disorder and compassion fatigue issues among emergency service nurses, this study is expected to make a significant contribution by identifying the level of earthquake trauma and compassion fatigue among nurses who experienced the 6 February Kahramanmaraş earthquakes and determining the relationship between them. The aim of this study is to determine the impact of earthquake trauma on compassion fatigue among nurses working in emergency services following the 6 February Kahramanmaraş earthquakes.

The following hypotheses will be tested within the scope of the research.

ELIGIBILITY:
Inclusion Criteria:

* Working in the emergency department of a hospital located in a province affected by the
* February 6 Kahramanmaraş earthquakes,
* Having worked in the emergency department for at least one year,
* Not having any psychiatric illness that could increase anxiety and stress levels in the last year,
* Not taking any medication that could affect anxiety and stress levels in the last year,
* Volunteering to participate in the study.

Exclusion Criteria:

* Data from nurses who wish to withdraw from the study after inclusion will not be considered for the research.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study targets emergency department nurses in areas affected by the February 6 Kahramanmaraş earthquakes in Turkey. These nurses, with at least one year of experience, have faced the disaster's challenges firsthand. The focus is on those actively involved in disaster response and recovery, excluding individuals with recent psychiatric conditions or medication that could influence stress levels. Participation is voluntary, ensuring data integrity and ethical standards. Nurses withdrawing from the study will have their data excluded.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Section 1: Demographic Information Form | up to 12 weeks
  This section of the data collection form includes questions aimed at identifying the nurses' age, gender, educational background, marital status, years of professional experience, years of experience in emergency services, monthly working hours after the earthquake, and work schedule (day, night, mixed). Additionally, this part contains questions regarding whether the nurses lost any relatives in the earthquake, the inhabitable damage to their homes, and if they were trapped under rubble. The Demographic Information Form consists of a total of 10 questions.
Section 2: Post-Earthquake Trauma Level Determination Scale | up to 12 weeks
  The Post-Earthquake Trauma Level Determination Scale (PETLDS) was developed by Tarhan and Hayri in 2013. The scale comprises 5 sub-dimensions: "Behavioral Problems," "Emotional Restriction," "Sensory Structuring," "Cognitive Structuring," and "Sleep Problems," consisting of a total of 20 negatively phrased items. Symptoms of post-traumatic stress are measured on a five-point Likert scale ranging from "strongly disagree" to "strongly agree." The lowest possible score on the scale is 20, and the highest is 100, with higher scores indicating a greater level of impact from the earthquake. Reliability analyses conducted by the creators resulted in Cronbach's alpha internal consistency coefficients of 0.64 for the first sub-dimension, 0.75 for the second, 0.61 for the third, 0.68 for the fourth, and 0.70 for the fifth. The overall internal consistency (Cronbach's alpha) for PETLDS was found to be 0.87. Cronbach's alpha will be recalculated with the research data.
Section 3: Compassion Fatigue Short Scale | up to 12 weeks
  Originally developed by Figley in 1995, this scale has a total of 13 items divided into two sub-dimensions: "Burnout" and "Secondary Traumatic Stress." In 2006, Adams et al. revised the scale, reducing it from 30 items to 13. The revision resulted in a Cronbach's alpha value of 0.90. The dimensions were redefined by Adams et al. as "Workload" and "Secondary Traumatic Stress," with Cronbach's alpha coefficients for these sub-dimensions found to be 0.80 and 0.90, respectively. Each item on the scale is scored from 1 to 10, with total scores ranging from 13 to 130; higher scores indicate higher levels of compassion fatigue. The Turkish adaptation of the scale was conducted by Yıldırım and Cavcav in 2020, confirming its validity and reliability in the Turkish population. The Cronbach's alpha value for the Turkish version was calculated as 0.91 by Yıldırım and Cavcav. The Cronbach's alpha for this research will be recalculated based on the research data.

CONTACTS AND LOCATIONS:
Overall Officials: islam elagöz, MsC, Study Director — devlet hastanesi
Locations (1):
- Islam Elagöz, Kilis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Informed Consent: Participants will be briefed about data sharing, including purposes and data types shared.
  De-identification: Data will be anonymized to remove personal identifiers, ensuring privacy.
  Data Repository: A secure platform will host the data, with access controlled through a data access request system.
  Data Use Agreement: Users must agree to use the data solely for research, adhere to data security protocols, and acknowledge the original study in publications.
  Monitoring: Compliance with the data use agreement will be monitored to prevent misuse.
  Timeframe: IPD will be available for a specified period after the study's main findings are published, with eventual secure archiving or destruction of the data.